CLINICAL TRIAL: NCT02040896
Title: Who Contributes to the Ordering of Computed Tomography in Emergency Department Patients? A Prospective Survey Study
Brief Title: Who Contributes to the Ordering of CT Scans in Emergency Department Patients?
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00047697
Record Dates: First submitted 2014-01-17; First posted 2014-01-20 (Estimated); Last update posted 2020-03-27 (Actual); Status verified 2020-01

CONDITIONS: Emergency
Keywords: computed tomography; emergency; CT scan; ordering behavior; diagnosis; radiation
MeSH Terms: conditions — Emergencies; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1: All consecutive emergency department patients undergoing CT during study hours will be prospectively enrolled, except for those meeting pre-specified exclusion criteria.

SUMMARY:
The primary objectives are:

1. To investigate which healthcare workers and other individuals contribute to the decision to order computed tomography (CT) scans for emergency department (ED) patients.
2. To investigate the specific reasons healthcare workers and other individuals order or request CT scans for ED patients.
3. To determine the frequency of clinically important actions following CT scan results.

Once the drivers of ED CT utilization are identified, interventions including education, incentives for compliance with evidence-based best practices, and interventions for noncompliance could be targeted appropriately.

ELIGIBILITY:
Inclusion Criteria:

- Patients from age 0 to <17 years, and patients age 18 years and older with traumatic and non-traumatic presentations, who visit Adult and Pediatric EDs and receive a CT scan during their ED visit

Exclusion Criteria:

* Patients older than 17, yet younger then 18.
* Patients who are unable to consent and who do not have a legally authorized representative.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients from age 0 to <17 years, and patients age 18 years and older with traumatic and non-traumatic presentations, who visit Adult and Pediatric EDs and receive a CT scan during their ED visit
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2014-01; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
CT scans utilization | January 2014 - January 2015
  Results will be categorized by body region of CT and patient age. For each CT region and age category, the percentage of CT scans requested by each demographic group (e.g., patient, emergency physician, etc.), will be reported, with 95% confidence intervals.
  CTs not requested by emergency physicians, the percentage of each type of scan requested by each demographic group will be reported, with 95% confidence intervals.

SECONDARY OUTCOMES:
Abnormal vs. normal CT scans | January 2014 - January 2015
  The frequency of abnormal CT results and clinical interventions will be calculated, for CTs requested by emergency physicians and for those not requested by emergency physicians (this includes all other parties).

CONTACTS AND LOCATIONS:
Overall Officials: Joshua S Broder, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Hospital, Durham, North Carolina, United States